CLINICAL TRIAL: NCT07169396
Title: Identification of Genetic Targets in Gynecological Tumors Via a Triple in Silico Ex-vivo / in Vivo Approach
Brief Title: Identifying Genetic Targets in Gynecological Tumors
Acronym: GEN_EXP_CO2021
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 676/2021/TESS/AUSLRE
Record Dates: First submitted 2025-08-29; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer
Keywords: gene expression; high-grade serous carcinoma; molecular oncology; tumor biomarkers
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Gene Expression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ovarian Cancer: Participants with high-grade serous ovarian carcinoma (HGSOC) or other rare epithelial ovarian tumor subtypes (e.g., mucinous, endometrioid, clear cell, mesonephric-like). Includes both prospectively enrolled patients and retrospectively collected samples. Purpose: to analyze gene and protein expression profiles in tumor tissues and compare them with normal ovarian epithelium.
  Interventions: Other: RNA extraction and gene expression
- Control group: Patients undergoing surgery for benign gynecological conditions, from whom non-tumoral ovarian epithelial tissue is obtained. Purpose: to provide baseline biological controls for comparison with ovarian cancer samples.
  Interventions: Other: RNA extraction and gene expression

INTERVENTIONS:
Other: RNA extraction and gene expression — RNA extraction and gene expression

SUMMARY:
This observational study aims to identfy genetic targets involved in the pathogenesis of gynecological tumors, with a focus on high-grade serous ovarian carcinoma. Using a triple approach - in silico, ex vivo and in vitro - the study will investigate the role of gonadotropins and their related signaling pathways in the epithelial ovarian cancers. Gene and protein expression levels will be evaluated through transcriptomic analysis, immunohistochemistry and functional assays on tumor cell lines. The goal is to uncover potential diagnostic or therapeutic targets in gynecological malignancies.

DETAILED DESCRIPTION:
Ovarian cancer is the leading cause of death among gynecological malignanciens. High-grade serous ovarian carcinoma (HGSOC) represents the most common and aggressive subtype. Growing evidence suggests that gonadotropins and their receptors (FSHR and LHCGR), as well as membrane estrogen receptors (GPER), may play a significant role in ovarian carcinogenesis by modulating proliferative and anti-apoptotic signals. The GEN EX CO 2021 study is a monocentric, observational project conducted at AUSL-IRCCS Reggio Emilia. It is both prospective and retrospective, and it aims to identify gene expression patterns that differentiate ovarian tumor tissues from normal ovarian epithelium. The study uses a triple experimental approach:

* In silico: differentially expressed genes were identified from public datasets (GSE18521 and GSE26712) via transcriptomic analysis and pathway analysis;
* Ex vivo: mRNA and protein expression will be assessed in fresh-frozen and FFPE tissue samples from patients with HGSOC and other rare epithelial ovarian tumor subtypes (e.g., mesonephric-like, mucinous, endometrioid, clear cell);
* In vitro: functional experiments using ovarian cancer cell lines (e.g., A2780, KGN, HGL5) will evaluate the effects of gene overexpression or silencing on cell viability, apoptosis and proliferation.

Participants include both prospective cases and retrospective samples, as well as control tissues from patients undergoing surgery for benign conditions. Gene expressions will be assessed through digital PCR, while protein levels will be analyzed via immunohistochemistry. Functional studies will explore the biological impact of selected genes on tumor cell behavior. Data will be collected using a secure, coded e-CRF in compliance with ethical and privacy regulations. The ultimate goal is to identify novel molecular targets that could inform future diagnostic or therapeutic approaches in ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult women ≥18 years old
* Histologically confirmed diagnosis of epithelial ovarian cancer (including high- grade serous, endometrioid, mucinous, clear cell, or mesonephric-like histotypes)
* Signed informed consent (for prospective cases) or ethically approved waiver (for retrospective samples)

Exclusion Criteria:

* Refusal to sign informed consent
* Diagnosis of low-grade or non-epithelial ovarian tumors
* Patients whose clinical or pathological data are unavailable or insufficient for study inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals assigned female at birth are eligible to participate in this study.
Study Population: Adult female patients diagnosed with epithelial ovarian cancer - including high-grade serous, endometrioid, mucinous, clear cell and mesonephric-like tumors - treated at AUSL-IRCCS Reggio Emilia, as well as women undergoing surgery for benign gynecological conditions (controls).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Gene expression profiling of selected target genes | 18 months
  Quantification of gene expression levels (e.g., PRKAR1A, GNAS, GNAQ, ERBB2, GPM6B, etc.) in ovarian tumor tissue vs normal ovarian epithelium using digital PCR.

SECONDARY OUTCOMES:
Protein expression analysis by immunohistochemistry | 24 months
  evaluation of protein levels of selected genes in ovarian tumor and control tissues.
Functional in vitro validation | 30 months
  assessment of cellular response to gene modulation (overexpression / silencing) in ovarian tumor cell lines.
Transcriptome-wide analysis in recurrent cases | 30 months
  extended differential gene expression and pathway analysis in samples from patients with tumor recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zheng W, Lu JJ, Luo F, Zheng Y, Feng Yj, Felix JC, Lauchlan SC, Pike MC. Ovarian epithelial tumor growth promotion by follicle-stimulating hormone and inhibition of the effect by luteinizing hormone. Gynecol Oncol. 2000 Jan;76(1):80-8. doi: 10.1006/gyno.1999.5628. PMID 10620446
- [Background] Zhang Z, Jia L, Feng Y, Zheng W. Overexpression of follicle-stimulating hormone receptor facilitates the development of ovarian epithelial cancer. Cancer Lett. 2009 Jun 8;278(1):56-64. doi: 10.1016/j.canlet.2008.12.024. Epub 2009 Jan 31. PMID 19181441
- [Background] Czogalla B, Partenheimer A, Jeschke U, von Schonfeldt V, Mayr D, Mahner S, Burges A, Simoni M, Melli B, Benevelli R, Bertini S, Casarini L, Trillsch F. beta-arrestin 2 Is a Prognostic Factor for Survival of Ovarian Cancer Patients Upregulating Cell Proliferation. Front Endocrinol (Lausanne). 2020 Sep 18;11:554733. doi: 10.3389/fendo.2020.554733. eCollection 2020. PMID 33042017
- [Background] Casarini L, Lazzaretti C, Paradiso E, Limoncella S, Riccetti L, Sperduti S, Melli B, Marcozzi S, Anzivino C, Sayers NS, Czapinski J, Brigante G, Poti F, La Marca A, De Pascali F, Reiter E, Falbo A, Daolio J, Villani MT, Lispi M, Orlando G, Klinger FG, Fanelli F, Rivero-Muller A, Hanyaloglu AC, Simoni M. Membrane Estrogen Receptor (GPER) and Follicle-Stimulating Hormone Receptor (FSHR) Heteromeric Complexes Promote Human Ovarian Follicle Survival. iScience. 2020 Nov 18;23(12):101812. doi: 10.1016/j.isci.2020.101812. eCollection 2020 Dec 18. PMID 33299978